CLINICAL TRIAL: NCT02855684
Title: 6-Month, Multicenter, Randomized, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® in Insulin-Naïve Patients With Type 2 Diabetes Mellitus Not Adequately Controlled With Non-Insulin Antihyperglycemic Drugs
Brief Title: Comparison of the Efficacy and Safety of a New Formulation of Insulin Glargine With Lantus in Patients With Type 2 Diabetes Insufficiently Controlled With Non-insulin Antidiabetic Therapy
Acronym: EDITION AP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12814; U1111-1139-3894 (Other: UTN)
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toujeo - insulin glargine (U300) (Experimental): Toujeo - Insulin glargine (U300) will be administered subcutaneously once in the evening on top of the non-insulin antihyperglycemic drugs for 29 weeks
  Interventions: Drug: Insulin glargine (U300); Drug: Non-insulin antihyperglycemic drugs
- Lantus - insulin glargine (Active Comparator): Lantus - Insulin glargine will be administered subcutaneously once in the evening on top of the non-insulin antihyperglycemic drugs for 29 weeks
  Interventions: Drug: Insulin glargine; Drug: Non-insulin antihyperglycemic drugs

INTERVENTIONS:
Drug: Insulin glargine (U300) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: HOE901; Toujeo
  Arms: Toujeo - insulin glargine (U300)
Drug: Insulin glargine — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: HOE901; Lantus
  Arms: Lantus - insulin glargine
Drug: Non-insulin antihyperglycemic drugs — Pharmaceutical form: capsule/tablet
  Route of administration: oral
  Other Names: Non-insulin antihyperglycemic therapy

SUMMARY:
Primary Objective:

To compare the efficacy of insulin glargine (U300) and Lantus in terms of change of glycated hemoglobin A1c (HbA1c) from baseline to endpoint (scheduled at Month 6, Week 26) in patients with type 2 diabetes mellitus.

Secondary Objectives:

* To compare insulin glargine (U300) and Lantus in terms of occurrence of hypoglycemia and nocturnal hypoglycemia.
* To compare insulin glargine (U300) and Lantus in terms of reaching target HbA1c values (all and reaching target without hypoglycemia).
* To compare insulin glargine (U300) and Lantus in terms of controlled plasma glucose (all and reaching target without hypoglycemia).
* To compare the frequency of occurrence and diurnal distribution of hypoglycemia by category of hypoglycemia (documented symptomatic, asymptomatic, nocturnal, severe, probable and relative).
* To assess the safety and tolerability of insulin glargine (U300).
* To assess the development of anti-insulin glargine antibodies (AIA).

DETAILED DESCRIPTION:
The total maximum study duration per patient will be 29 weeks that will consist of a 2-week screening period, 26-week treatment period, and a 2-day post-treatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Adult patients with type 2 diabetes mellitus inadequately controlled with non-insulin antihyperglycemic drug(s).
* Signed written informed consent.

Exclusion criteria:

* Age < legal age of adulthood.
* HbA1c <7.0% (<53 mmol/mol) or >11% (>97 mmol/mol) (at screening).
* History of type 2 diabetes mellitus for less than 1 year before screening.
* Less than 6 months before screening with non-insulin antihyperglycemic treatment.
* Change in dose of non-insulin antihyperglycemic treatment in the last 3 month before screening.
* Initiation of new glucose-lowering medications and/or weight loss drug in the last 3 months before screening visit and/or initiation of glucagon like peptide-1(GLP-1) receptor agonist in the last 6 months before screening visit.
* Patients receiving only non-insulin antihyperglycemic drugs not approved for combination with insulin according to local labeling (Note: non-insulin antihyperglycemic drugs not approved for combination with insulin are to be discontinued at randomization).
* Current or previous insulin use except for a maximum of 10 consecutive days (eg, acute illness, surgery) during the last one year prior to screening.
* Severe hypoglycemia resulting in coma/seizures, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eg, laser, surgical treatment or injectable drugs) during the study period.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2016-08-24; Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | Baseline, 6 months

SECONDARY OUTCOMES:
Percentage (%) of patients with at least one hypoglycemia | Baseline, up to 6 months
Percentage (%) of patients with at least one nocturnal hypoglycemia | Baseline, up to 6 months
Percentage (%) of patients with HbA1c <7.0% | 6 months
Percentage (%) of patients with HbA1c ≤6.5% | 6 months
Percentage (%) of patients with Fasting Plasma Glucose (FPG) <100 mg/dL (5.6 mmol/L) | 6 months
Percentage (%) of patients with FPG ≤120 mg/dL (6.7 mmol/L) | 6 months
Percentage (%) of patients requiring rescue therapy | 6 months
Change in fasting plasma glucose | Baseline, 6 months
Change in 8-point Self-monitored Plasma Glucose (SMPG) profiles | Baseline, 6 months
Change of mean 24-hour plasma glucose | Baseline, 6 months
Change in variability of plasma glucose profile | Baseline, 6 months
Change in daily basal insulin dose | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (54):
- China (39):
  - Investigational Site Number 1560039, Beijing
  - Investigational Site Number 1560001, Beijing
  - Investigational Site Number 1560017, Beijing
  - Investigational Site Number 1560003, Beijing
  - Investigational Site Number 1560033, Changchun
  - Investigational Site Number 1560016, Changzhou
  - Investigational Site Number 1560049, Changzhou
  - Investigational Site Number 1560006, Fuzhou
  - Investigational Site Number 1560004, Guangzhou
  - Investigational Site Number 1560036, Guangzhou
  - Investigational Site Number 1560043, Guangzhou
  - Investigational Site Number 1560014, Guangzhou
  - Investigational Site Number 1560042, Guiyang
  - Investigational Site Number 1560024, Hangzhou
  - Investigational Site Number 1560046, Hefei
  - Investigational Site Number 1560025, Hohhot
  - Investigational Site Number 1560019, Jinan
  - Investigational Site Number 1560027, Lanzhou
  - Investigational Site Number 1560038, Nanchang
  - Investigational Site Number 1560045, Nanchang
  - Investigational Site Number 1560002, Nanjing
  - Investigational Site Number 1560012, Nanjing
  - Investigational Site Number 1560047, Nanjing
  - Investigational Site Number 1560021, Shanghai
  - Investigational Site Number 1560018, Shanghai
  - Investigational Site Number 1560048, Shenyang
  - Investigational Site Number 1560005, Shenyang
  - Investigational Site Number 1560020, Shenzhen
  - Investigational Site Number 1560013, Siping
  - Investigational Site Number 1560031, Tangshan
  - Investigational Site Number 1560023, Tianjin
  - Investigational Site Number 1560044, Tianjin
  - Investigational Site Number 1560009, Xi'an
  - Investigational Site Number 1560034, Xiamen
  - Investigational Site Number 1560010, Xuzhou
  - Investigational Site Number 1560026, Yueyang
  - Investigational Site Number 1560011, Zhengzhou
  - Investigational Site Number 1560030, Zhenjiang
  - Investigational Site Number 1560041, Zhuzhou
- South Korea (11):
  - Investigational Site Number 4100003, Anyang
  - Investigational Site Number 4100005, Busan
  - Investigational Site Number 4100010, Gwangju
  - Investigational Site Number 4100012, Gyeonggi-do
  - Investigational Site Number 4100008, Seoul
  - Investigational Site Number 4100001, Seoul
  - Investigational Site Number 4100009, Seoul
  - Investigational Site Number 4100004, Seoul
  - Investigational Site Number 4100006, Seoul
  - Investigational Site Number 4100007, Seoul
  - Investigational Site Number 4100002, Wŏnju
- Taiwan (4):
  - Investigational Site Number 1580001, Taichung
  - Investigational Site Number 1580004, Taipei
  - Investigational Site Number 1580003, Taipei
  - Investigational Site Number 1580002, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org